CLINICAL TRIAL: NCT00955474
Title: The Efficacy and Tolerability of Seroquel XR Combined With a Selective Serotonin Re-Uptake Inhibitor Versus Seroquel XR Monotherapy in the Acute Treatment of Major Depressive Disorder With Psychotic Features
Brief Title: Seroquel Alone Versus Seroquel With an SSRI for Depression With Psychotic Symptoms
Acronym: Seroquel
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: AstraZeneca halted funding; patent expired for Seroquel (Quetiapine) in 2012
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, John D. Matthews, Director of Inpatient Research & Training, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008P001022
Record Dates: First submitted 2009-08-06; First posted 2009-08-10 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Major Depressive Disorder With Psychotic Features
MeSH Terms: interventions — Quetiapine Fumarate; Escitalopram; Sertraline; Citalopram

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quetiapine (Experimental): Patients assigned to receive Quetiapine
  Interventions: Drug: Quetiapine
- Quetiapine and SSRI (Active Comparator): Patients assigned to receive Quetiapine and SSRI
  Interventions: Drug: Quetiapine; Drug: escitalopram; Drug: Sertraline; Drug: Citalopram

INTERVENTIONS:
Drug: Quetiapine — Quetiapine XR 100 mg/h.s. will be the starting dose and increased by 100 mg q h.s. q day to a target dose of 300 mg/h.s. by day three and continued on 300 mg/h.s. through week three. Between weeks four and eight, there will be flexible dosing up to 800 mg/h.s. or reductions in doses to no lower than 200 mg/h.s. Incremental increases or decreases in dose will be no more than 100 mg/h.s. over a minimum of one week, unless a patient is unable to tolerate the current dose. Patients unable to tolerate at least 200 mg/h.s. will be discontinued from the study.
  Other Names: Quetiapine (generic name): Seroquel (brand name)
Drug: escitalopram — Active comparator arm:
  Escitalopram 5 mg/a.m. starting dose; increase to 10 mg/a.m. at week 2 and continued at 10 mg/a.m. through week 3. Weeks 4-8: flexible dosing up to 20 mg/a.m. or reductions in doses to no lower than 5 mg/a.m.
  Other Names: Lexapro
  Arms: Quetiapine and SSRI
Drug: Sertraline — Active comparator arm:
  Sertraline 50 mg/a.m. starting dose; increased to 100 mg/a.m. at week 2; continued on 100 mg/a.m. through week 3. Weeks 4-8: flexible dosing up to 200 mg/a.m. or reductions in doses to no lower than 50 mg/a.m.
  Citalopram 20 mg/a.m. starting dose; increased to a target dose of 40 mg/a.m. at week 2; continued on 40 mg/a.m. through Week 8: reductions in doses to no lower than 20 mg/a.m.
  Escitalopram 5 mg/a.m. starting dose; increase to 10 mg/a.m. at week 2 and continued at 10 mg/a.m. through week 3. Weeks 4-8: flexible dosing up to 20 mg/a.m. or reductions in doses to no lower than 5 mg/a.m.
  Other Names: Zoloft (brand name)
  Arms: Quetiapine and SSRI
Drug: Citalopram — Active comparator arm:
  Citalopram 20 mg/a.m. starting dose; increased to a target dose of 40 mg/a.m. at week 2; continued on 40 mg/a.m. through Week 8: reductions in doses to no lower than 20 mg/a.m.
  Other Names: Celexa
  Arms: Quetiapine and SSRI

SUMMARY:
The purpose of this study is to compare the efficacy and tolerability of Seroquel monotherapy for the treatment of Major Depression with Psychotic features with Seroquel plus Selective Serotonin Reuptake Inhibitor.

DETAILED DESCRIPTION:
The proposed study is designed to investigate the non-inferiority of treatment of PsyD using monotherapy with quetiapine XR versus combination treatment using quetiapine XR and an SSRI (sertraline or citalopram or escitalopram) during the acute phase of treatment. The primary outcome measures will be the change rates of symptoms of depression (as measured on the Hamilton Rating Scale for Depression [HAM-D-17] and psychosis (as measured on the Brief Psychiatric Rating Scale [BPRS] Positive Symptoms Subscale).

The secondary aim of the study is to assess the safety and efficacy of the combination of quetiapine XR and SSRIs in patients with the diagnosis of PsyD. Metabolic factors including fasting glucose, fasting insulin, and fasting lipids (total cholesterol, HDL, LDL, and triglycerides) will be obtained at screen and at the 8-week endpoint of the study to assess the impact of treatment on the development of risk factors for metabolic syndrome. Measures of cognitive function (MGH Cognitive and Physical Functioning Questionnaire and RBANS) (Fava et al. 2006; Randolph et al. 1998) will be obtained at screen and the 8-week endpoint of the study to assess the impact of treatment on cognitive function.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Diagnosis of Major Depressive Disorder with Psychotic Features by the DSM-IV
3. Females and Males between the ages of 18-85 years.
4. Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrolment
5. Able to understand and comply with the requirements of the study
6. Initial HAM-D-17 score of > 16, both at the screen visit and at the baseline visit.
7. Participants must have an initial BPRS score of > 25 and at least one of the following: > 5 for item 1, > 5 for item 5, > 5 for item 8, > 4 for item 9, > 1 for item 10, > 1 for item 11; these BPRS criteria msut be met both at the screen visit and at the baseline visit.
8. Participants must have an initial CGI score of > 2, both at the screen visit and at the baseline visit.

Exclusion Criteria:

1. Pregnancy or lactation
2. Any DSM-IV Axis I disorder not defined in the inclusion criteria
3. Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
4. Known intolerance or lack of response to quetiapine fumarate, as judged by the investigator
5. Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
6. Use of any of the following cytochrome P450 inducers in the 14 days preceding enrollment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
7. Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomization
8. Substance or alcohol dependence within the past three months (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria
9. Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrolment
10. Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
11. Unstable or inadequately treated medical illness (e.g. diabetes, angina pectoris, hypertension) as judged by the investigator
12. Involvement in the planning and conduct of the study
13. Previous enrolment or randomization of treatment in the present study.
14. Participation in another drug trial within 4 weeks prior enrollment into this study or longer in accordance with local requirements
15. A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria:

    * Unstable DM defined as enrollment glycosylated hemoglobin (HbA1c) > 8.5%.
    * Admitted to hospital for treatment of DM or DM related illness in past 12 weeks.
    * Not under physician care for DM.
    * Physician responsible for patient's DM care has not indicated that patient's DM is controlled.
    * Physician responsible for patient's DM care has not approved patient's participation in the study
    * Has not been on the same dose of oral hypoglycaemic drug(s) and/or diet for the 4 weeks prior to randomization. For thiazolidinediones (glitazones) this period should not be less than 8 Weeks.
    * Taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks
16. An absolute neutrophil count (ANC) of 1.5 x 10^9 per liter
17. Patients with a history seizure disorder; unstable physical disorders (cardiovascular, hepatic, renal, respiratory, endocrine, neurologic, or hematologic); or any physical disorder judged to significantly affect central nervous system function.
18. Patients who are currently treated with antidepressants other than the selective serotonin reuptake inhibitors, with mood stabilizing or antipsychotic drugs other than quetiapine.
19. Patients with known arrhythmias or arrhythmias noted on screening EKG.
20. Outpatients with a CGI score of 7.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D Matthews, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruitment through newspaper advertisements in the Boston metro area.
Pre-assignment Details: Participants were required to wash-out prior to randomization and study procedures. If the patient was unable to wash-out (by personal choice or doctor's recommendation), they were excluded. Seven subjects withdrew consent prior to randomization.
Groups:
- Quetiapine: Patients assigned to receive Quetiapine
  •Quetiapine XR 100 mg/h.s. will be the starting dose and increased by 100 mg q h.s. q day to a target dose of 300 mg/h.s. by day three and continued on 300 mg/h.s. through week three. Between weeks four and eight, there will be flexible dosing up to 800 mg/h.s. or reductions in doses to no lower than 200 mg/h.s. Incremental increases or decreases in dose will be no more than 100 mg/h.s. over a minimum of one week, unless a patient is unable to tolerate the current dose. Patients unable to tolerate at least 200 mg/h.s. will be discontinued from the study.
- Quetiapine and SSRI: Patients assigned to receive Quetiapine and SSRI
  * Quetiapine XR 100 mg/h.s. starting dose; increased by 100 mg q h.s. q day; target dose 300 mg/h.s. by day 3; continued on 300 mg/h.s. through week 3. Weeks 4-8: flexible dosing up to 800 mg/h.s. or reductions in doses to no lower than 200 mg/h.s.
  * Sertraline 50 mg/a.m. starting dose; increased to 100 mg/a.m. at week 2; continued on 100 mg/a.m. through week 3. Weeks 4-8: flexible dosing up to 200 mg/a.m. or reductions in doses to no lower than 50 mg/a.m.
  * Citalopram 20 mg/a.m. starting dose; increased to a target dose of 40 mg/a.m. at week 2; continued on 40 mg/a.m. through Week 8: reductions in doses to no lower than 20 mg/a.m.
  * Escitalopram 5 mg/a.m. starting dose; increase to 10 mg/a.m. at week 2 and continued at 10 mg/a.m. through week 3. Weeks 4-8: flexible dosing up to 20 mg/a.m. or reductions in doses to no lower than 5 mg/a.m.
Period: Overall Study
Arm/Group | Quetiapine | Quetiapine and SSRI
Started | 12 | 13
Completed | 5 | 8
Not Completed | 7 | 5
Not completed — Physician Decision | 7 | 5

BASELINE CHARACTERISTICS:
Population: Thirty-two patients were consented and 25 participants were randomized. The remaining 7 participants withdrew consent prior to randomization and the collection of any baseline data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Quetiapine | Quetiapine and SSRI | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 13 | 25
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 39.25 [25 to 58] | 42.85 [21 to 62] | 40.32 [21 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 8 | 9 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 8 | 12 | 20
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 9 | 8 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Depression
Description: Depression measured with Hamilton Rating Scale for Depression 17 (HAM-D) at baseline and 8 weeks. Ham D 17 scores range from 0-52, 52 being the most severe.
Time Frame: 8 weeks
Population: Missing data for two subjects in the quetiapine with SSRI group;11 of 13 have baseline outcome measures. There were five completers (8 weeks) in the quetiapine group and 8 completers (8 weeks) in the quetiapine with SSRI group.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Quetiapine With SSRI: Patients assigned to receive Quetiapine and SSRI
  * Quetiapine XR 100 mg/h.s. starting dose; increased by 100 mg q h.s. q day; target dose 300 mg/h.s. by day 3; continued on 300 mg/h.s. through week 3. Weeks 4-8: flexible dosing up to 800 mg/h.s. or reductions in doses to no lower than 200 mg/h.s.
  * Sertraline 50 mg/a.m. starting dose; increased to 100 mg/a.m. at week 2; continued on 100 mg/a.m. through week 3. Weeks 4-8: flexible dosing up to 200 mg/a.m. or reductions in doses to no lower than 50 mg/a.m.
  * Citalopram 20 mg/a.m. starting dose; increased to a target dose of 40 mg/a.m. at week 2; continued on 40 mg/a.m. through Week 8: reductions in doses to no lower than 20 mg/a.m.
  * Escitalopram 5 mg/a.m. starting dose; increase to 10 mg/a.m. at week 2 and continued at 10 mg/a.m. through week 3. Weeks 4-8: flexible dosing up to 20 mg/a.m. or reductions in doses to no lower than 5 mg/a.m.
Arm/Group | Quetiapine | Quetiapine With SSRI
Number analyzed (Participants) | 12 | 11
units on a scale
  Baseline | 27 (16.21) | 26.73 (6.84)
  Last visit: number analyzed (Participants) | 5 | 8
  Last visit | 9.57 (5.44) | 10.14 (8.40)

2. Primary Outcome: Psychosis
Description: Psychosis measured by Brief Psychosis Rating Scale (BPRS) at baseline and 8 weeks. Scores range from 24-168, with 168 bring the most severe.
Time Frame: 8 weeks
Population: Complete missing data for 2 subjects in the quetiapine with SSRI group (11 of 13 have baseline outcome measures). There were 5 completers (8 weeks) in the quetiapine group and 8 completers (8 weeks) in the quetiapine with SSRI group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine | Quetiapine With SSRI
Number analyzed (Participants) | 12 | 11
units on a scale
  Baseline | 56.09 (7.26) | 60.45 (16.49)
  Last visit: number analyzed (Participants) | 5 | 8
  Last visit | 34.25 (25.04) | 32.83 (8.98)

3. Secondary Outcome: Fasting Blood Glucose
Description: Fasting glucose levels collected at Baseline and Week 8. Normal range for fasting glucose is 70-110 mg/dl.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ml/dl
Arm/Group | Quetiapine | Quetiapine and SSRI
Number analyzed (Participants) | 12 | 11
ml/dl
  Baseline | 91.6 (10.2) | 89.4 (10.6)
  Week 8: number analyzed (Participants) | 5 | 8
  Week 8 | 89.1 (2.2) | 96.8 (19.2)

4. Secondary Outcome: CPFQ (Cognitive and Psychological Functioning Questionnaire)
Description: Score on the Cognitive and Psychological Functioning Questionnaire (CPFQ). Scores range from 7-42 with 42 referring to the worst functioning. CPFQ measured at baseline and 8 weeks.
Time Frame: 8 weeks
Population: Missing data for two subjects in the quetiapine with SSRI group;11 of 13 have baseline outcome measures. There were 5 completers (8 weeks) in the quetiapine group and 8 completers (8 weeks) in the quetiapine with SSRI group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine | Quetiapine With SSRI
Number analyzed (Participants) | 12 | 11
units on a scale
  Baseline | 30.8 (4.69) | 29.3 (9.24)
  Last visit: number analyzed (Participants) | 5 | 8
  Last visit | 23.56 (7.07) | 21.00 (6.40)

5. Secondary Outcome: RBANS (Repeatable Battery for Assessment of Neuropsychological Status) Total Score
Description: Neuropsychological Assessment. Scores range from 40-160, with 160 referring to higher cognitive functioning. All RBANS subscales and the total score are standardized using age-based norms. Thus, they have a mean of 100 (average) and a standard deviation of 15. A score of 90-110 is in the average range; score of 70-85 mild to moderate cognitive impairment; score <70 moderate to severe impairment. RBANS measured at baseline and 8 weeks.
Time Frame: 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine | Quetiapine With SSRI
Number analyzed (Participants) | 12 | 11
units on a scale
  Baseline | 77.38 (13.71) | 70.00 (16.12)
  Last visit: number analyzed (Participants) | 5 | 8
  Last visit | 77.25 (15.23) | 78.29 (16.94)

6. Secondary Outcome: RBANS (Repeatable Battery for Assessment of Neuropsychological Status) Immediate Memory Sub-scale Score
Description: RBANS Immediate Memory sub-scale scores at Baseline and Week 8. Scores range from 40-160, with 160 referring to higher cognitive functioning. All RBANS subscales and the total score are standardized using age-based norms. Thus, they have a mean of 100 (average) and a standard deviation of 15. A score of 90-110 is in the average range; score of 70-85 mild to moderate cognitive impairment; score <70 moderate to severe impairment.
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine | Quetiapine With SSRI
Number analyzed (Participants) | 12 | 11
units on a scale
  Baseline | 83.3 (17.2) | 71.1 (14.1)
  Week 8: number analyzed (Participants) | 5 | 8
  Week 8 | 82.8 (14.4) | 77.9 (16.2)

7. Secondary Outcome: RBANS (Repeatable Battery for Assessment of Neuropsychological Status) Visuospatial/Constructional Sub-scale.
Description: RBANS Visuospatial/Constructional sub-scales at Baseline and Week 8. Scores range from 40-160, with 160 referring to higher cognitive functioning. All RBANS subscales and the total score are standardized using age-based norms. Thus, they have a mean of 100 (average) and a standard deviation of 15. A score of 90-110 is in the average range; score of 70-85 mild to moderate cognitive impairment; score <70 moderate to severe impairment.
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine | Quetiapine With SSRI
Number analyzed (Participants) | 12 | 11
units on a scale
  Baseline | 70.6 (15.9) | 75.6 (16.1)
  Week 8: number analyzed (Participants) | 5 | 8
  Week 8 | 70.5 (30.8) | 78.3 (17.8)

8. Secondary Outcome: RBANS (Repeatable Battery for Assessment of Neuropsychological Status) Language Sub-scale Score.
Description: RBANS Language sub-scale scores at Baseline and Week 8 of study. Scores range from 40-160, with 160 referring to higher cognitive functioning. All RBANS subscales and the total score are standardized using age-based norms. Thus, they have a mean of 100 (average) and a standard deviation of 15. A score of 90-110 is in the average range; score of 70-85 mild to moderate cognitive impairment; score <70 moderate to severe impairment.
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine | Quetiapine With SSRI
Number analyzed (Participants) | 12 | 11
units on a scale
  Baseline | 80.4 (16.2) | 77.6 (21.2)
  Week 8: number analyzed (Participants) | 5 | 8
  Week 8 | 87.9 (13.7) | 91.1 (7.9)

9. Secondary Outcome: RBANS (Repeatable Battery for Assessment of Neuropsychological Status) Attention Sub-scale Scores at Baseline and Week 8.
Description: RBANS Attention sub-scale scores at Baseline and Week 8. Scores range from 40-160, with 160 referring to higher cognitive functioning. All RBANS subscales and the total score are standardized using age-based norms. Thus, they have a mean of 100 (average) and a standard deviation of 15. A score of 90-110 is in the average range; score of 70-85 mild to moderate cognitive impairment; score <70 moderate to severe impairment.
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine | Quetiapine With SSRI
Number analyzed (Participants) | 12 | 11
units on a scale
  Baseline | 95.8 (17.1) | 85.4 (15.9)
  Week 8: number analyzed (Participants) | 5 | 8
  Week 8 | 104.6 (21.6) | 86.1 (11.0)

10. Secondary Outcome: RBANS (Repeatable Battery for Assessment of Neuropsychological Status) Delayed Memory Subscale Scores at Baseline and Week 8.
Description: RBANS Delayed Memory subscale scores at Baseline and Week 8. Scores range from 40-160, with 160 referring to higher cognitive functioning. All RBANS subscales and the total score are standardized using age-based norms. Thus, they have a mean of 100 (average) and a standard deviation of 15. A score of 90-110 is in the average range; score of 70-85 mild to moderate cognitive impairment; score <70 moderate to severe impairment.
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine | Quetiapine With SSRI
Number analyzed (Participants) | 12 | 11
units on a scale
  Baseline | 82.4 (21.6) | 69.6 (22.3)
  Week 8: number analyzed (Participants) | 5 | 8
  Week 8 | 72.9 (13.7) | 74.7 (24.3)

11. Secondary Outcome: Blood Level of Total Cholesterol Levels Were Collected at Baseline and Week 8.
Description: Cholesterol levels were collected at Baseline and Week 8. Normal cholesterol levels should be <200mg/dl.
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Quetiapine | Quetiapine With SSRI
Number analyzed (Participants) | 12 | 11
mg/dl
  Baseline | 184.2 (34.4) | 171.8 (38.8)
  Week 8: number analyzed (Participants) | 5 | 8
  Week 8 | 188 (2.2) | 201.7 (55.8)

12. Secondary Outcome: Blood Level of Triglycerides at Baseline and Week 8.
Description: Level of triglycerides at Baseline and Week 8. Normal range: 40-150mg/dl.
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Quetiapine | Quetiapine With SSRI
Number analyzed (Participants) | 12 | 11
mg/dl
  Baseline | 144.9 (71.1) | 154.25 (80.5)
  Week 8: number analyzed (Participants) | 5 | 8
  Week 8 | 170.6 (125.2) | 190.5 (68.5)

13. Secondary Outcome: HDL Blood Levels at Baseline and Week 8.
Description: HDL levels at Baseline and Week 8. Normal range: 35-100 mg/dl.
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Quetiapine | Quetiapine With SSRI
Number analyzed (Participants) | 12 | 11
mg/dl
  Baseline | 47.7 (15.1) | 45.3 (6.6)
  Week 8: number analyzed (Participants) | 5 | 8
  Week 8 | 40.8 (13.2) | 40.5 (12.2)

14. Secondary Outcome: LDL Blood Levels at Baseline and Week 8.
Description: LDL levels at Baseline and Week 8. Normal range < 100 mg/dl.
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Quetiapine | Quetiapine With SSRI
Number analyzed (Participants) | 12 | 11
mg/dl
  Baseline | 109 (25.3) | 94.6 (27.3)
  Week 8: number analyzed (Participants) | 5 | 8
  Week 8 | 121.1 (39.4) | 123.3 (42.2)

15. Secondary Outcome: Blood Hemoglobin A1C at Baseline and Week 8.
Description: Blood hemoglobin A1C at Baseline and Week 8. Normal range: 3.8%-6.4%.
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: % glycated hemoglobin
Arm/Group | Quetiapine | Quetiapine With SSRI
Number analyzed (Participants) | 12 | 11
% glycated hemoglobin
  Baseline | 5.6 (0.5) | 5.7 (0.5)
  Week 8: number analyzed (Participants) | 5 | 8
  Week 8 | 5.4 (0.5) | 5.8 (0.3)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Quetiapine | Quetiapine and SSRI
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 2/12 | 1/13
Other Adverse Events (participants affected / at risk) | 8/12 | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quetiapine (N=12) | Quetiapine and SSRI (N=13)
Acute mania (Nervous system disorders) | 0 | 1 — The patient was hospitalized for acute mania and it was considered unrelated.
Worsening depression (Psychiatric disorders) | 1 (1) | 0 (0) — Severity of depression resulted in psychiatric hospitalization. Considered to be unrelated to the study.
Increased paranoia and auditory hallucinations (Psychiatric disorders) | 1 (1) | 0 (0) — The worsening psychosis resulted in psychiatric hospitalization.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quetiapine (N=12) | Quetiapine and SSRI (N=13)
Excess sedation (Psychiatric disorders) | 2 (2) | 4 (4) — Sedation is a common side effect from Seroquel
Leg cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Fatigue (Nervous system disorders) | 2 (2) | 5 (5)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dreaming (Psychiatric disorders) | 0 (0) | 1 (1)
Headaches (Nervous system disorders) | 0 (0) | 1 (1)
Light headedness (Cardiac disorders) | 1 (1) | 1 (1)
Dry mouth (Nervous system disorders) | 3 (3) | 2 (2)
Hand weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sweating (Nervous system disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Carbohydrate cravings (Nervous system disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No